CLINICAL TRIAL: NCT07406841
Title: Comparison of Spinal and General Anesthesia on Maternal and Neonatal Outcomes in Pregnancies With Placenta Accreta Spectrum: A Retrospective Study
Brief Title: Spinal Versus General Anesthesia in Pregnancies With Placenta Accreta Spectrum: A Retrospective Comparative Study
Acronym: SAGA-PAS
Status: Not yet recruiting | Type: Observational
Sponsor: Gaziantep City Hospital (Other)
Responsible Party: Principal Investigator, Recep Karakaşoğlu, Principal Investigator, Gaziantep City Hospital
Other Study IDs: GZŞH-ANES-PAS-2025
Record Dates: First submitted 2026-02-03; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Placenta Accreta Spectrum
Keywords: Placenta accreta spectrum; PAS; spinal anesthesia; general anesthesia
MeSH Terms: conditions — Placenta Accreta | interventions — Anesthesia, Spinal; Anesthesia, General

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Spinal Anesthesia: This cohort includes pregnant patients diagnosed with placenta accreta spectrum who underwent cesarean delivery under spinal anesthesia as part of routine clinical care. The anesthetic technique was selected by the multidisciplinary clinical team based on standard institutional practice and individual patient characteristics. No experimental intervention was applied for research purposes.
  Interventions: Procedure: spinal anesthesia
- General Anesthesia: This cohort includes pregnant patients diagnosed with placenta accreta spectrum who underwent cesarean delivery under general anesthesia as part of routine clinical care. The anesthetic technique was selected by the multidisciplinary clinical team based on standard institutional practice and individual patient characteristics. No experimental intervention was applied for research purposes.
  Interventions: Procedure: General Anesthesia

INTERVENTIONS:
Procedure: spinal anesthesia — Spinal anesthesia administered for cesarean delivery as part of routine clinical care in pregnant patients with placenta accreta spectrum. The technique was chosen by the clinical team based on standard institutional practice and patient condition, not for research assignment.
  Groups: Spinal Anesthesia
Procedure: General Anesthesia — General anesthesia was administered for cesarean delivery in pregnant patients with placenta accreta spectrum as part of routine clinical care. The anesthetic technique, including airway management, induction agents, and maintenance strategy, was selected by the attending anesthesia team according to institutional standards and the patient's clinical condition. The intervention was not assigned for research purposes.
  Groups: General Anesthesia

SUMMARY:
Placenta accreta spectrum (PAS) is a serious pregnancy complication in which the placenta grows abnormally into the uterine wall. This condition is associated with a high risk of severe bleeding, need for blood transfusion, hysterectomy, and maternal complications during cesarean delivery.

This study aims to compare spinal anesthesia and general anesthesia in pregnant women diagnosed with placenta accreta spectrum who underwent cesarean delivery. The researchers reviewed existing medical records to evaluate differences in maternal and neonatal outcomes between the two anesthesia approaches.

The primary outcomes include changes in hemoglobin levels before and after surgery, the need for uterotonic medications during and after the operation, and newborn Apgar scores. Because this is a retrospective observational study, no new treatments were given, and all data were collected from routine clinical care records.

The findings are expected to help guide anesthetic decision-making in PAS cases, improve maternal and neonatal safety, and contribute to the international scientific literature on this topic.

DETAILED DESCRIPTION:
This is a single-center, retrospective observational study conducted in pregnant patients diagnosed with placenta accreta spectrum (PAS) who underwent cesarean delivery at Gaziantep City Hospital. Medical records were reviewed to identify eligible cases between the predefined study period based on imaging findings, intraoperative diagnosis, and/or histopathological confirmation of PAS.

Patients were categorized according to the type of anesthesia received during cesarean delivery: spinal anesthesia or general anesthesia. The choice of anesthetic technique was based on routine clinical practice, multidisciplinary team decision, and individual patient characteristics, rather than random assignment. No additional interventions were introduced for research purposes.

Data were extracted from electronic medical records, anesthesia charts, obstetric files, and neonatal records. Collected variables included demographic characteristics, obstetric history, imaging findings suggestive of PAS, intraoperative management strategies, estimated blood loss, transfusion requirements, use of uterotonic agents, and perioperative hemodynamic parameters. Neonatal data included gestational age at delivery, birth weight, Apgar scores at 1 and 5 minutes, need for resuscitation, and admission to neonatal intensive care.

The primary analytic focus was the comparison of perioperative hemoglobin change between the spinal and general anesthesia groups. Secondary analyses evaluated differences in intraoperative and postoperative uterotonic requirements, transfusion needs, surgical complications, length of hospital stay, and neonatal outcomes.

Statistical analyses were performed using appropriate parametric or non-parametric tests depending on data distribution. Potential confounding factors such as placenta previa status, prior cesarean history, and PAS severity were considered in subgroup analyses.

Ethics approval was obtained from the Gaziantep City Hospital Clinical Research Ethics Committee prior to data collection, and patient confidentiality was maintained in accordance with national regulations and the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant patients diagnosed with placenta accreta spectrum (PAS), Undergoing elective cesarean delivery, Receiving either spinal anesthesia or general anesthesia during cesarean section, Singleton pregnancy, Availability of complete medical and anesthesia records related to surgery and perioperative management

Exclusion Criteria:

Patients without a diagnosis of PAS, Emergency (non-elective) cesarean deliveries, Use of anesthesia techniques other than spinal or general anesthesia, Multiple pregnancy (twins or more) ,Incomplete or missing medical/anesthesia records, Missing key perioperative or neonatal outcome data

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population consists of pregnant women diagnosed with placenta accreta spectrum (PAS) who underwent elective cesarean delivery at Gaziantep City Hospital. Participants were identified retrospectively from hospital medical records and anesthesia charts. Only patients with singleton pregnancies and complete perioperative and neonatal data were included in the analysis. The population reflects routine clinical practice in the management of PAS at a tertiary care center.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-02-01 (Actual); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Length of Hospital Stay to Discharge | Postoperative day of hospital discharge, assessed up to 30 days after cesarean delivery.
  Total duration of maternal hospitalization calculated from the time of cesarean delivery until official hospital discharge.
Perioperative Hemoglobin Change | From preoperative assessment to 48 hours after cesarean delivery
  The difference between preoperative hemoglobin level and postoperative hemoglobin level measured within the first 48 hours after cesarean delivery in patients with placenta accreta spectrum.
Neonatal Apgar Score at 1 and 5 Minutes | At 1 minute and 5 minutes after birth
  Neonatal Apgar scores assessed at 1 and 5 minutes after birth in infants delivered by cesarean section in pregnancies with placenta accreta spectrum.